CLINICAL TRIAL: NCT03580018
Title: Intraarticular Injection of Tranexamic Acid Reduced Postoperative Hemarthrosis in Arthroscopic Anterior Cruciate Ligament Reconstruction - A Prospective Randomized Study
Brief Title: Intraarticular Injection of Tranexamic Acid Reduced Postoperative Hemarthrosis in Arthroscopic Anterior Cruciate Ligament Reconstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-07-004B
Record Dates: First submitted 2018-06-26; First posted 2018-07-09 (Actual); Last update posted 2018-07-12 (Actual); Status verified 2018-07

CONDITIONS: Anterior Cruciate Ligament Reconstruction
Keywords: Anterior cruciate ligament reconstruction, knee, hemarthrosis, tranexamic acid
MeSH Terms: conditions — Hemarthrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tranexamic Acid group (Experimental): Ten mL of TXA (100 mg/mL) was injected into the joint at the end of the index operation and the drain was clamped for 2 h.
  Interventions: Drug: Tranexamic Acid Powder
- Control Group (Placebo Comparator): The control group patients only received ACLRs without TXA injections.
  Interventions: Procedure: Post-anterior cruciate ligament reconstruction (ACLR)

INTERVENTIONS:
Drug: Tranexamic Acid Powder — Ten mL of Tranexamic Acid(100 mg/mL) was injected into the joint at the end of the operation.
  Arms: Tranexamic Acid group
Procedure: Post-anterior cruciate ligament reconstruction (ACLR) — Post-anterior cruciate ligament reconstruction (ACLR)
  Arms: Control Group

SUMMARY:
Post-anterior cruciate ligament reconstruction (ACLR) hemarthrosis may result in increased pain thus delaying postoperative rehabilitation, which may eventually lead to arthrofibrosis and a functional deficit. Many antifibrinolytic agents, including tranexamic acid (TXA), have been used in orthopedic surgeries to reduce postoperative bleeding.The purpose of this study is to evaluate the effect of intra-articular injection of TXA in patients receiving arthroscopic ACLRs. Patients were randomized into two groups. Group 1 patients (TXA group) received the index procedures with a 10 mL intra-articular injection of TXA. Group 2 (control group) patients received the index procedures without TXA injections. An intra-articular suction drain was placed recorded 24 h postoperatively. Clinical evaluations using an IKDC functional score, range of motion (ROM), and a Visual Analogue Scale (VAS) pain score were performed at postoperative day 3 and week 4.

DETAILED DESCRIPTION:
TXA group patients received ACLRs and a 10 mL intra-articular injection of TXA after the procedure. The control group patients only received ACLRs without TXA injections. Randomization was done on the day of the surgery, by an independent investigator who did not participate in the surgery, using the permuted block randomization technique.

The same surgeon treated all patients enrolled in this study. Spinal anesthesia was given to all patients and a pneumatic tourniquet was routinely used. In brief, through a 3 cm incision over the medial proximal tibia, semitendinosus (ST) and gracilis (Gr) tendons were harvested from the distal insertion. Tendons were quadrupled and whip stitched by No. 2 and No. 5 Ethibond sutures (Ethicon, Somerville, NJ). The diameters of the folded tendons were determined by using sizing cylinders with incremental size changes of 0.5 mm.The femoral sockets were created at about the 1:30 position (left knee), through the anteromedial portal. The tibial tunnel was created with an ACUFEX guide (Smith & Nephew, Andover, MA). The diameters of the socket were created in the same manner as the diameter of the folded graft. At tibial site, grafts were fixed with bioscrews (BIORCI-HA, Smith & Nephew) at 30 degrees of knee flexion. The screw and the tunnel sizes were the same. After completion of the procedure, a suction drain (Zimmer HEMOVAC, Warsaw, IN) was placed at the superior lateral aspect of the joint. Ten mL of TXA (100 mg/mL) (Daiichi Sankyo, Tokyo, Japan) was injected into the joint at the end of the operation and the drain was clamped for 2 h.

Clinical evaluations The volume of drainage was recorded 24 h after surgery. The grade of hemarthrosis, as previously described by Coupens et al.,was also documented at day 3 and week The range of knee motion and the IKDC functional score were evaluated 4 weeks post-surgery. The VAS was documented at postoperative day 3 and week 4.

Statistical analysis. All data are expressed as a mean and standard deviation (SD). The amount of drainage or functional scores between different groups were compared with an independent t test.

All statistical analyses were conducted using SPSS version 11.0 (SPSS Inc., Chicago,IL). Differences were considered significant when the p-value was < 0.05.

ELIGIBILITY:
Inclusion Criteria:

1. patient agreed to participate in this study, signed an informed consent document.
2. patients receiving arthroscopic ACLR with autologous hamstring grafts

Exclusion Criteria:

1. previous knee procedures on the same side
2. renal disorder or insufficiency
3. abnormal coagulation profile
4. refused to participate in this study

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 320 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
The volume of drainage | 24 hours after surgery.
  hemoarthrosis

SECONDARY OUTCOMES:
The grade of hemarthrosis | At day 3 and week 4.
  Grade I to IV.
The VAS was documented | Postoperative day 3 and week 4.
  scale 0 to 10.
IKDC functional score | Evaluated 4 weeks post-surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Hsiao-Li, Taipei, Taiwan